CLINICAL TRIAL: NCT05339256
Title: A Randomized, Controlled Trial of Sublingual Buprenorphine Through Telemedicine vs In-Person Care as Usual in the Treatment of Opioid Use Disorder
Brief Title: Sublingual Buprenorphine Through Telemedicine vs In-Person Care as Usual
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Christina Ann Brezing, Assistant Professor of Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8305; R21DA055835 (NIH)
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: randomized, active-control, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Telehealth buprenorphine induction and maintenance (Experimental): Sublingual (SL) Buprenorphine and a medical management protocol adapted to the unique needs of home-based telehealth for MOUD using SL buprenorphine
  Interventions: Drug: Buprenorphine SL; Other: Telehealth
- Standard in-person SL buprenorphine induction and maintenance (Active Comparator): In-person induction and maintenance dosing of sublingual buprenorphine, or MOUD as usual.
  Interventions: Drug: Buprenorphine SL; Other: In-person treatment as usual

INTERVENTIONS:
Drug: Buprenorphine SL — Up to 24 mg per day
Other: Telehealth — Telehealth MOUD, utilizing a standardized protocol for each healthcare provider session
  Arms: Telehealth buprenorphine induction and maintenance
Other: In-person treatment as usual — in-person induction and maintenance dosing of sublingual buprenorphine, or MOUD as usual.
  Arms: Standard in-person SL buprenorphine induction and maintenance

SUMMARY:
This study will compare in-person induction and maintenance dosing of sublingual buprenorphine to induction and maintenance dosing of sublingual buprenorphine through comprehensive telehealth sessions and telehealth medication for opioid use disorder (MOUD).

DETAILED DESCRIPTION:
The study is a 12-week, randomized, active-control, open-label, early phase II effectiveness trial of telemedicine treatment using sublingual buprenorphine as compared to in person clinic treatment with sublingual buprenorphine for outpatients seeking treatment for opioid use disorder (OUD). This telehealth protocol serves as a model of the integration of evidence-based practices in medication for opioid use disorder (MOUD) and could be used by non addiction specialists at scale. The primary outcome will be time to dropout. Participants will have daily study visits (either in person or remote) during the initial buprenorphine induction week and then twice per week during the maintenance phase (either in person or remote) over the 12-week trial. Remote visits will be conducted using the HIPAA-compliant technology, FaceTime and/or Webex.

ELIGIBILITY:
Inclusion Criteria:

* meet DSM-5 criteria for OUD
* Voluntarily seeking buprenorphine treatment for OUD
* Able to provide informed consent and comply with study procedures

Exclusion Criteria:

* Meeting DSM-5 criteria for substance use disorder other than opioid as the primary diagnosis that would compromise safety of participation in the trial as determined by the study physician, such as an alcohol or sedative hypnotic use disorder that requires detoxification
* Having a comorbid psychiatric diagnosis that might interfere with participation or make participation hazardous, such as a psychotic disorder including schizophrenia or schizoaffective disorder
* Concurrent methadone, buprenorphine, or vivitrol maintenance treatment
* Known history of allergy, intolerance, or hypersensitivity to candidate medication (buprenorphine)
* Pregnancy, lactation, or failure to use adequate contraceptive methods in female patients
* Unstable medical conditions, such as severe hepatic, renal, or cardiovascular disease, which might make participation
* Current or recent history history of significant violent or suicidal behavior or risk for suicide or homicide
* Legally mandated to substance use disorder treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to drop out | 12 weeks
  Comparing time to drop out between the treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Christina Brezing, MD, Principal Investigator — New York State Psychiatric Institute

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published in this report (after de-identification) (text, tables, figures)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning twelve months and ending 5 years after article publication
Access Criteria: to researcher who provides a methodologically sound proposal to achieve aims in approved proposal